CLINICAL TRIAL: NCT03250390
Title: Analysis of Volatile Organic Compounds in Exhaled Air as a Diagnostic Tool for Thoracic Cancers
Brief Title: Breath Analysis to Diagnose Lung Cancer
Acronym: CATOCOV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Institut National de Recherche en Informatique et en Automatique (Other); Institut Pasteur de Lille (Other); Institut MinesTelecom (IMT) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017_05; 2017-A00932-51 (Other: ID-RCB Number, ANSM); PHRCI_2016 (Other: PHRC number,DGOS)
Record Dates: First submitted 2017-08-07; First posted 2017-08-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Lung Cancer
Keywords: Lung cancer; diagnosis; volatile organic compounds
MeSH Terms: conditions — Lung Neoplasms; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients (Experimental): Patients with bronchopulmonary cancer who have not yet received therapeutic treatment.
  Interventions: Device: Collection of volatile organic compounds during exhalation
- controls (Active Comparator): The controls consisted of 2 groups: smokers and non-smokers.
  Interventions: Device: Collection of volatile organic compounds during exhalation

INTERVENTIONS:
Device: Collection of volatile organic compounds during exhalation — The volatile organic compounds (VOCs) are collected in sorbents at rest and at the end of exhalation according to the concentration of carbon dioxide using ReCIVA breath sampler.
  The identification of the VOCs will be done by chromatography (Gas Chromatography Mass Spectrometry GC-MS)

SUMMARY:
Determination of volatile organic compounds to discriminate patients with lung cancer from healthy smokers and non-smokers healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* patients with histologically proven lung cancer

Controls:

* healthy smoker or non-smoker subjects
* without respiratory diseases excepted chronic obstructive pulmonary disease.

Exclusion Criteria:

* history of cancer other than lung cancer within 5 years before inclusion
* oral or facial malformation
* incomprehension of maneuvers for the collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Actual)
Dates: Start 2019-04-29 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2024-04-29 (Actual)

PRIMARY OUTCOMES:
Discriminating power of VOCs | 34 months
  Discriminating power of VOCs using discriminant analyzes using innovative data mining methods based on multi-objective combinatorial optimization.

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien Hulo, MD, Principal Investigator — University Hospital, Lille
Locations (7):
- France (7):
  - Institut Pasteur - Centre de Prévention et d'Education à la Santé (CPES), Lille
  - Hôpital Calmette, CHU, Lille
  - Hopital Victor Provo, Roubaix
  - Centre Hospitalier de Saint Quentin, Saint-Quentin
  - Chu Amiens Salouël, Salouël
  - Ch Seclin - Seclin, Seclin
  - Clinique Teissier, Valenciennes

IPD SHARING:
Plan to Share IPD: No